CLINICAL TRIAL: NCT04335305
Title: A Randomized, Controlled, Open-Label, Phase II Trial to Evaluate the Efficacy and Safety of Tocilizumab Combined With Pembrolizumab (MK-3475) in Patients With Coronavirus Disease 2019 (COVID-19)-Pneumonia
Brief Title: Checkpoint Blockade in COVID-19 Pandemic
Acronym: COPERNICO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP376; 2020-001160-28 (EudraCT Number)
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — tocilizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab plus Pembrolizumab (MK-3475) (Experimental): Tocilizumab 8 mg/kg (up to a maximum of 800 mg per dose) as an intravenous infusion over 60 minutes; single dose Pembrolizumab (MK3475) 200 mg as an intravenous infusion over 30 minutes; single dose.
  Patients who are showing no clinical improvement in respiratory function after 12 hours could receive an additional dose of tocilizumab at the same dose level of the first administration. Patients who are showing SpO2 ≤ 94% on room air could receive an additional administration of pembrolizumab (MK-3475) at the same recommended dose after 3 weeks from treatment initiation and/or an additional dose of tocilizumab after 4 weeks from treatment initiation at physician's discretion.
  Interventions: Drug: Tocilizumab; Biological: Pembrolizumab (MK-3475)
- Continued Standard of Care (No Intervention): Standard care per local written policies or guidelines comprises, as necessary and at physician's discretion, supplemental oxygen, noninvasive and invasive ventilation, antibiotic agents, vasopressor support, renal-replacement therapy, glucocorticoid, tocilizumab, virally targeted agents, chloroquine or hydroxychloroquine.

INTERVENTIONS:
Drug: Tocilizumab — IV infusion over 60 minutes; 8 mg/kg (up to a maximum of 800 mg per dose); single dose
  Other Names: Actemra; RoActemra
  Arms: Tocilizumab plus Pembrolizumab (MK-3475)
Biological: Pembrolizumab (MK-3475) — IV infusion over 30 minutes, 200 mg; single dose
  Other Names: MK-3475; Keytruda
  Arms: Tocilizumab plus Pembrolizumab (MK-3475)

SUMMARY:
This is a prospective, multicenter, randomized, controlled, open-label, phase 2 clinical trial

DETAILED DESCRIPTION:
The aim of this study is to assess the efficacy -as determined by the proportion of patients with normalization of SpO2 ≥96% on room air- of continued standard care together with tocilizumab plus pembrolizumab (MK- 3475) in patients with COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form (ICF) prior to participation in any study-related activities.

   Note: If no written ICF can be provided by the trial participant, consent could be given either orally in the presence of an impartial witness or from the legal representative in accordance with national and local patient regulations.
2. Male or non-pregnant female patients ≥ 18 years and ≤ 80 years at the time of ICF.
3. Laboratory confirmed COVID-19 infection defined with a positive reverse transcription-polymerase chain reaction (RT-PCR) from any specimen and/or detection of SARS-CoV-2 immunoglobulin (Ig)M/IgG antibodies.
4. Diagnostic confirmation of pneumonia by either chest X-ray or thoracic CT scan (preferable).
5. Patient with acute respiratory syndrome related to COVID-19.
6. Patients with Sequential Organ Failure Assessment (SOFA) score ≤ 3 at the time of ICF.
7. Patients with total lymphocyte count ≤0,8 x106/mL.
8. Patients who are showing SpO2 ≤ 92% on room air (measured without any respiratory support for at least 15 minutes). Note: For patients on prior tocilizumab-containing regimen, SpO2 ≤ 94% on room air is sufficient criterion for their eligibility.
9. Patients who meet at least one of the following parameters: • Increased levels of ferritin;

   * Increased levels of IL-6;
   * Increased levels of D-dimer;
   * Increased levels of CRP;
   * Increased levels of LDH;
   * Increased levels of ESR;
   * For patients on prior tocilizumab-containing regimen for COVID-19, no objective clinical improvement at physician's discretion within 48 hours after treatment initiation.
10. Life expectancy greater than 10 days.
11. Willing to take study medication and to comply with all study procedures.
12. In women of childbearing potential, negative pregnancy test and commitment to use contraceptive method throughout the study.

Exclusion criteria

1. Participation in any other clinical trial of an experimental treatment for COVID-19.
2. Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 is prohibited < 24 hours prior to study drug dosing, except the commonly used antiviral drugs and/or chloroquine and/or tocilizumab.
3. Requiring endotracheal intubation, mechanical ventilation, and extracorporeal membrane oxygenation (ECMO) at screening.
4. Patients being treated with immunomodulators or anti-rejection drugs.
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN).
6. Creatinine clearance < 50 mL/min.
7. Chronic Obstructive Pulmonary Disease (COPD) or end-stage lung disease that require home oxygen therapy.
8. Known hypersensitivity to recombinant proteins, or any excipient contained in the drug formulation of study pembrolizumab and tocilizumab.
9. Treatment with high doses of systemic corticosteroids within 72 hours prior obtaining consent except for inhaled steroids and prior corticosteroid therapy at dose lower than or equal to 10 mg/day methylprednisolone equivalent.
10. Bowel diverticulitis or perforation.
11. Diagnosis of immunodeficiency receiving immunosuppressive therapy within seven days prior to study treatment initiation. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
12. Current known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if PCR test is negative for HCV ribonucleic acid (RNA).
13. Vaccination with any live virus vaccine within 28 days prior to study treatment initiation.

    Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live-attenuated vaccines and are not allowed.
14. History of prior allogeneic bone marrow, stem-cell, or solid organ transplantation.
15. Patients have any other concurrent severe medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.
16. Pregnant women, lactating women and planned pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with normalization of SpO2 ≥96% on room air (measured without any respiratory support for at least 15 minutes | through day 14 after study treatment initiation
  Assessed by hospital records

SECONDARY OUTCOMES:
Proportion of patients discharged from the emergency department and classified as low risk | through End of Study, defined as 90 ± 14 days after study entry
  Assessed by hospital records
Number of days of patient hospitalization | through End of Study, defined as 90 ± 14 days after study entry
  Assessed by hospital records
Change from baseline in organ failure parameters | Days 1, 3, 5, 7, 14 (+/- 1 day) and 28 (+/- 2 days) or until discharge whatever it comes first.
  The clinical status will be assessed by the SOFA scores
Proportion of mortality rate | through End of Study, defined as 90 ± 14 days after study entry
  Determined as percentage of dead patients
Analysis of the remission of respiratory symptoms | through End of Study, defined as 90 ± 14 days after study entry
  Determined as:
  * Time to invasive mechanical ventilation (if not previously initiated);
  * Time to independence from non-invasive mechanical ventilation;
  * Time to independence from oxygen therapy.
Evaluation of the radiological response | at days 1 and 28 (+/- 2 days)
  by using the same imaging technique (chest X-ray or thoracic CT scan)
Time to first negative in severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) RT-PCR test | within 28 days from study inclusion
  determined using oropharyngeal or anal swabs
Change from baseline of absolute lymphocyte count (ALC),white blood cell count and white blood cell differential count | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of hemoglobin | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of platelets | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of activated partial thromboplastin time (aPTT) | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of creatinine | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of glucose | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of total bilirubin | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Change from baseline of albumin | days 3, 5, 7, 10, 14 and 28 after administration of study drug
  Baseline defined as the value collected at day 1, 2 hours before treatment administration
Incidence of adverse events (AEs), incidence of prespecified AEs (safety and tolerability) | Up to End of Study, defined as 90 ± 14 days after study entry
  Evaluated using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v.5.0), SOFA scores.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, Study Chair — IOB Institute of Oncology, Vall d´Hebron Institute of Oncology (VHIO)
Locations (7):
- Spain (7):
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Ruber Juan Bravo, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Arnau de Vilanova-Lliria, Valencia
  - Hospital Universitario Doctor Peset, Valencia